CLINICAL TRIAL: NCT03135574
Title: Prevalence of a High-intensity Signal of the Oculomotor Nerve on T2 MRI Sequence in Patients With Ophthalmoplegia
Acronym: HYPER-III
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: FHN_2016_27
Record Dates: First submitted 2017-04-25; First posted 2017-05-01 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Ophthalmoplegia
MeSH Terms: conditions — Ophthalmoplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI T2 sequence of the oculomotor tract — Patients with ophthalmoplegia will benefit from an MRI T2 sequence of the oculomotor tract (additional time of 4 minutes).

SUMMARY:
Oculomotor nerve (third cranial nerve or III) palsy is a relatively frequent cause of consultation in ophthalmology.

It may reveal a life-threatening pathology such as aneurysm rupture, pituitary apoplexy, and therefore need imaging in emergency. Apart from few extreme emergency situations, MRI of the oculomotor tract is the first-line examination required. In the usual clinical practice, the investigators noticed in several patients unusual areas of high-intensity signal within the oculomotor nerve on T2 sequence, observed in various locations along the nerve path (cavernous and/ or intra-orbital segment). This abnormal signal, at the best knowledge of the investigators, has never been reported in the literature and could confirm the nerve impairment.

In patients with ophthalmoplegia involving probably the third cranial nerve, disclosing this new MRI sign could help (i) to confirm the involvement of the oculomotor nerve and eliminate differential diagnoses such as myasthenia (ii) to orientate the etiological diagnosis (inflammatory or ischemic origin). A T2 sequence focused on the III could thus be systematically included in the usual MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

* Ophthalmoplegia whatever the clinical form (unilateral or not, isolated or not, sudden or progressive onset)

Exclusion Criteria:

* Absolute contraindication to MRI or injection of contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (18 years of age or older) benefiting from an MRI, requested by the ophthalmologist for an assessment of an ophthalmoplegia.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-04-16 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
High-intensity signal of the oculomotor nerve on MRI T2 sequence (presence or absence, determined by a radiologist) | Baseline
  High-intensity signal within the oculomotor nerve on T2 sequence, observed in various locations along the nerve path (cavernous and/ or intra-orbital segment).
  High-intensity signal on T2 MRI sequence is defined as a signal area which is more intense than the contralateral nerve or more intense than the white matter signal.
  A double separate reading of the imaging will be carried out by an experienced radiologist and a junior radiologist on anonymized MRIs, with no access to clinical elements and interpretation of the other radiologist. In case of discrepancy between the radiologists, the final decision will be made by a third experienced radiologist under the same conditions (no access to clinical data, no access to the other evaluations).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France